CLINICAL TRIAL: NCT00005181
Title: Blood Pressure Control in Juveniles - Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1059; R01HL035795 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To correlate dietary factors and changes in pressor substances, including aldosterone and norepinephrine, with blood pressure during growth and sexual development from childhood through adolescence.

DETAILED DESCRIPTION:
BACKGROUND:

Blood pressure increases with age, and over time, reaches proportions consistent with clinically defined hypertension in some individuals. The age-dependent increase in blood pressure starts in mid-childhood and accelerates during puberty and in the post-pubertal period. Thus, mechanisms for the development of hypertension are likely present at an early age. The National Heart, Lung, and Blood Institute sponsored the 'Workshop on Juvenile Hypertension' in May 1983. The Workshop conclusions were that although a great deal had been accomplished in the past decade, research in juvenile hypertension had slowed and little effort was evident in some important areas of the field. They noted especially the paucity of effort in research relating to mechanisms of blood pressure regulation and elevation, to clinical management of the hypertensive state, and to identification of the prehypertensive state. Based on the recommendations of the Workshop, this study was initiated in response to a Request for Applications on 'Juvenile Hypertension and the Prehypertensive State' released by the NHLBI in October 1984.

DESIGN NARRATIVE:

Production of aldosterone and norepinephrine is examined in a mixed-longitudinal study design in white and Black boys and girls beginning at ages 6 to 12 and extending to age 17. Levels of these pressor systems are determined in the basal state from measurements made in urine samples collected overnight. To enhance the likelihood that school children would comply with the multiple observations required for this longitudinal study, measurements are deliberately restricted to non-invasive ones. Specifically, aldosterone and norepinephrine excretion measured in sleep urine are obtained at six month intervals in addition to blood pressure, heart rate, weight, height, and skin-fold thickness. Family history of hypertension and parental blood pressures are used as covariates in analysis of data in children. A second part of the study concerns the observation that blood pressure increases at a faster rate during adrenarche, a period of increasing adrenal androgen production, and during puberty. Androgen production during periods of adrenal and gonadal maturation may contribute to the increase in blood pressure. The relationship of androgen to blood pressure is examined by distinguishing blood pressure responses to androgen production from effects of androgens on physical growth, thus exploring the concept that androgens interact directly with pressor systems to raise blood pressure. Androgen production during the adrenarche is determined by measurement of dehydroepiandrosterone-sulfate excretion, and during puberty by measurement of luteinizing hormone excretion in sleep urine samples. Studies continue on the relationship between aldosterone excretion rate, dietary potassium intake, and blood pressure. A cross-over study is conducted to examine the effect of potassium supplementation on aldosterone production. Segregation analysis of the 'low-aldosterone'phenotype is performed on family members of children with low-aldosterone.

The study was renewed in 1996 to continue the longitudinal study of children (a biracial population, ages 6-16 years) for whom influences of hormones on blood pressure are being examined. Twice yearly the children have had blood pressure and anthropometrics measured, and overnight urine samples collected for measurement of aldosterone, adrenal androgens (AA), luteinizing hormone (LH), sodium, potassium, and creatinine. Rates of growth and the changes in blood pressure with age have been well characterized for this population. From the original observations, several differences were observed between racial groups; specifically, Black children were found to consume less potassium, produce about 40 percent less aldosterone and have higher blood pressures than white children. It was observed that children with positive families histories of hypertension were more likely to have lower aldosterone-excretion rates.

As part of the proposed continuation of longitudinal studies, the hypothesis is tested that children with low-aldosterone levels are predisposed to higher blood pressures. Although Black children had lower potassium intakes, cross-sectional data indicated that only part of the racial difference in aldosterone production was secondary to a lower intake of potassium (potassium is a known stimulus of aldosterone production). Subjects with known low-aldosterone production (Blacks and whites) have diets supplemented with potassium to test the hypothesis that Blacks with low-aldosterone production have a reduced responsiveness to potassium when compared to white children with low-aldosterone. Families of children with potassium-resistant low-aldosterone production are screened for evidence of low-aldosterone production, and segregation analyses is performed to establish the mode of inheritance of the 'low-aldosterone' phenotype. In cross-sectional studies, AA-excretion rates were positively related to blood pressure in subjects greater than or equal to 10 years of age, suggesting an important role for the adrenarche in determining blood pressure levels in young people. In future longitudinal studies the role of AA as well as gonadal hormones will be studied as more children reach adolescence (the current mean age of the cohort is 12.7 yr). In addition, to better distinguish the individual influences of adrenarche, gonadarche, and increases in body size on blood pressure, a series of patients where these phenomenon are dissociated will be studied.

The study was renewed in FY 2002 to identify new mechanisms for hypertension using a strategy which identifies the sodium transporters in kidney that account for why blacks retain more sodium than whites. Three sites along the nephron will be studied based on compelling evidence that they are linked to the increased sodium-retention in blacks.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pratt — Indiana University School of Medicine

REFERENCES:
- [Background] Bloem LJ, Foroud TM, Ambrosius WT, Hanna MP, Tewksbury DA, Pratt JH. Association of the angiotensinogen gene to serum angiotensinogen in blacks and whites. Hypertension. 1997 May;29(5):1078-82. doi: 10.1161/01.hyp.29.5.1078. PMID 9149669
- [Background] Pratt JH, Manatunga AK, Hanna MP, Ambrosius WT. Effect of administered potassium on the renin-aldosterone axis in young blacks compared with whites. J Hypertens. 1997 Aug;15(8):877-83. doi: 10.1097/00004872-199715080-00012. PMID 9280211
- [Background] Pratt JH, Jones JJ, Miller JZ, Wagner MA, Fineberg NS. Racial differences in aldosterone excretion and plasma aldosterone concentrations in children. N Engl J Med. 1989 Oct 26;321(17):1152-7. doi: 10.1056/NEJM198910263211703. PMID 2677724
- [Background] Pratt JH, Manatunga AK, Wagner MA, Jones JJ, Meaney FJ. Adrenal androgen excretion during adrenarche. Relation to race and blood pressure. Hypertension. 1990 Oct;16(4):462-7. doi: 10.1161/01.hyp.16.4.462. PMID 2145221
- [Background] Pratt JH, Manatunga AK, Bowsher RR, Henry DP. The interaction of norepinephrine excretion with blood pressure and race in children. J Hypertens. 1992 Jan;10(1):93-6. doi: 10.1097/00004872-199201000-00015. PMID 1312558
- [Background] Manatunga AK, Reister TK, Miller JZ, Pratt JH. Genetic influences on the urinary excretion of aldosterone in children. Hypertension. 1992 Feb;19(2):192-7. doi: 10.1161/01.hyp.19.2.192. PMID 1737654
- [Background] Pratt JH, Rothrock JK, Dominguez JH. Inhibition of aldosterone production by pinacidil in vitro. Hypertension. 1991 Oct;18(4):529-34. doi: 10.1161/01.hyp.18.4.529. PMID 1655650
- [Background] Shackleton CH, Kletke C, Wudy S, Pratt JH. Dehydroepiandrosterone sulfate quantification in serum using high-performance liquid chromatography/mass spectrometry and a deuterated internal standard: a technique suitable for routine use or as a reference method. Steroids. 1990 Oct;55(10):472-8. doi: 10.1016/0039-128x(90)90016-5. PMID 2149221
- [Background] Pratt JH, Manatunga AK, Peacock M. A comparison of the urinary excretion of bone resorptive products in white and black children. J Lab Clin Med. 1996 Jan;127(1):67-70. doi: 10.1016/s0022-2143(96)90167-5. PMID 8592098
- [Background] Bloem LJ, Manatunga AK, Pratt JH. Racial difference in the relationship of an angiotensin I-converting enzyme gene polymorphism to serum angiotensin I-converting enzyme activity. Hypertension. 1996 Jan;27(1):62-6. doi: 10.1161/01.hyp.27.1.62. PMID 8591889
- [Background] Bloem LJ, Guo C, Pratt JH. Identification of a splice variant of the rat and human mineralocorticoid receptor genes. J Steroid Biochem Mol Biol. 1995 Nov;55(2):159-62. doi: 10.1016/0960-0760(95)00162-s. PMID 7495694
- [Background] Bloem LJ, Manatunga AK, Tewksbury DA, Pratt JH. The serum angiotensinogen concentration and variants of the angiotensinogen gene in white and black children. J Clin Invest. 1995 Mar;95(3):948-53. doi: 10.1172/JCI117803. PMID 7883995
- [Background] Pratt JH, Manatunga AK, Li W. Familial influences on the adrenal androgen excretion rate during the adrenarche. Metabolism. 1994 Feb;43(2):186-9. doi: 10.1016/0026-0495(94)90243-7. PMID 8121300
- [Background] Pratt JH, Manatunga AK, Bloem LJ, Li W. Racial differences in aldosterone excretion: a longitudinal study in children. J Clin Endocrinol Metab. 1993 Dec;77(6):1512-5. doi: 10.1210/jcem.77.6.8263135.
- [Background] Manatunga AK, Jones JJ, Pratt JH. Longitudinal assessment of blood pressures in black and white children. Hypertension. 1993 Jul;22(1):84-9. doi: 10.1161/01.hyp.22.1.84. PMID 8319996
- [Background] Pratt JH, Ambrosius WT, Tewksbury DA, Wagner MA, Zhou L, Hanna MP. Serum angiotensinogen concentration in relation to gonadal hormones, body size, and genotype in growing young people. Hypertension. 1998 Nov;32(5):875-9. doi: 10.1161/01.hyp.32.5.875. PMID 9822447
- [Background] Ambrosius WT, Compton JA, Bowsher RR, Pratt JH. Relation of race, age, and sex hormone differences to serum leptin concentrations in children and adolescents. Horm Res. 1998;49(5):240-6. doi: 10.1159/000023178. PMID 9568809
- [Background] Zhou L, Ambrosius WT, Newman SA, Wagner MA, Pratt JH. Heart rate as a predictor of future blood pressure in schoolchildren. Am J Hypertens. 2000 Oct;13(10):1082-7. doi: 10.1016/s0895-7061(00)00295-8. PMID 11041162
- [Background] Jakubowski H, Ambrosius WT, Pratt JH. Genetic determinants of homocysteine thiolactonase activity in humans: implications for atherosclerosis. FEBS Lett. 2001 Feb 23;491(1-2):35-9. doi: 10.1016/s0014-5793(01)02143-3. PMID 11226414
- [Background] Ambrosius WT, Newman SA, Pratt JH. Rates of change in measures of body size vary by ethnicity and gender. Ethn Dis. 2001 Spring-Summer;11(2):303-10. PMID 11456005
- [Background] Pratt JH, Ambrosius WT, Agarwal R, Eckert GJ, Newman S. Racial difference in the activity of the amiloride-sensitive epithelial sodium channel. Hypertension. 2002 Dec;40(6):903-8. doi: 10.1161/01.hyp.0000039749.75068.f4. PMID 12468577
- [Background] Pratt JH, Eckert GJ, Newman S, Ambrosius WT. Blood pressure responses to small doses of amiloride and spironolactone in normotensive subjects. Hypertension. 2001 Nov;38(5):1124-9. doi: 10.1161/hy1101.095010. PMID 11711509
- [Background] Degawa-Yamauchi M, Dilts JR, Bovenkerk JE, Saha C, Pratt JH, Considine RV. Lower serum adiponectin levels in African-American boys. Obes Res. 2003 Nov;11(11):1384-90. doi: 10.1038/oby.2003.187. PMID 14627760
- [Background] Palacios C, Wigertz K, Martin BR, Jackman L, Pratt JH, Peacock M, McCabe G, Weaver CM. Sodium retention in black and white female adolescents in response to salt intake. J Clin Endocrinol Metab. 2004 Apr;89(4):1858-63. doi: 10.1210/jc.2003-031446. PMID 15070956
- [Background] Chun TY, Pratt JH. Non-genomic effects of aldosterone: new actions and questions. Trends Endocrinol Metab. 2004 Oct;15(8):353-4. doi: 10.1016/j.tem.2004.08.002. PMID 15380805
- [Background] Shankar RR, Ferrari P, Dick B, Ambrosius WT, Eckert GJ, Pratt JH. Activity of 11beta-hydroxysteroid dehydrogenase type 2 in normotensive blacks and whites. Ethn Dis. 2005 Summer;15(3):407-10. PMID 16108299
- [Background] Saha C, Eckert GJ, Pratt JH, Shankar RR. Onset of overweight during childhood and adolescence in relation to race and sex. J Clin Endocrinol Metab. 2005 May;90(5):2648-52. doi: 10.1210/jc.2004-2208. Epub 2005 Feb 22. PMID 15728215
- [Background] Shankar RR, Eckert GJ, Saha C, Tu W, Pratt JH. The change in blood pressure during pubertal growth. J Clin Endocrinol Metab. 2005 Jan;90(1):163-7. doi: 10.1210/jc.2004-0926. Epub 2004 Oct 27. PMID 15509638